CLINICAL TRIAL: NCT05786781
Title: An Exploratory Study on the Application of Transarterial CT Angiography in the Interventional Treatment of Massive Hemoptysis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UHCT22759
Record Dates: First submitted 2023-02-20; First posted 2023-03-28 (Actual); Last update posted 2025-04-13 (Actual); Status verified 2025-04

CONDITIONS: Hemoptysis
MeSH Terms: conditions — Hemoptysis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Transarterial CT angiography (Experimental): Transarterial catheter-directed CT angiography during interventional treatment of hemoptysis
  Interventions: Device: Transarterial CT angiography

INTERVENTIONS:
Device: Transarterial CT angiography — Transarterial catheter-directed CT angiography during interventional treatment of hemoptysis

SUMMARY:
This is a single-arm, exploratory study to evaluate the value of transarterial CT angiography applying Nexaris Angio-CT in the interventional treatment of massive hemoptysis

ELIGIBILITY:
Inclusion Criteria:

* Patients with massive hemoptysis（defined as more than 100mL per session or more than 300mL/day or with acute respiratory failure requiring mechanical ventilation or hemodynamic instability (systolic blood pressure < 90 mmHg), regardless of hemoptysis amount）

Exclusion Criteria:

* Pregnancy
* Patients with a previous history of bronchial artery embolization
* Uncorrectable severe infection, coagulation dysfunction, organ failure or cachexia, severe contrast agent allergy, and other interventional treatment contraindications

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2023-03-28 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
The accuracy rate of transarterial CT angiography in the identification of culprit vessel | Intraoperative phase
  The accuracy rate of transarterial CT angiography in the identification of culprit vessel, by calculating the matching rate between Angio-CT and selective angiography findings.
In-hospital clinical success | During the postoperative hospitalization period (i.e., the period after bronchial artery embolization until discharge)
  either the complete cessation of hemoptysis or a clinically significant reduction in bleeding, defined as ≤ 5 mL/24 hours of blood-tinged sputum or fresh blood during the hospitalization period.
Early hemoptysis recurrence rate | 3 months after treatment
  Recurrence rate of hemoptysis within 3 months after treatment

SECONDARY OUTCOMES:
Technical success rate | Intraoperative phase
  Technical success is defined as complete cessation of target blood flow confirmed by DSA
Radiation exposure | Intraoperative phase
  Radiation exposure data were systematically collected from structured radiation dose reports. For Angio-CT scans, radiation exposure was quantified using the volume CT dose index (CTDIvol) and dose-length product (DLP). For digital subtraction angiography (DSA) and fluoroscopy, air kerma (AK) and dose-area product (DAP) were utilized as metrics.
The amount of contrast agent consumed | Intraoperative phase
  The amount of contrast agent consumed during treatment
Adverse events | Intraoperative phase and during 3 months after treatment
  AEs were monitored and classified according to the Common Terminology Criteria for Adverse Events (CTCAE), version 5.0. The CTCAE system grades AEs on a 5-point scale, with grade ≥ 3 denoting a serious AE.

CONTACTS AND LOCATIONS:
Locations (1):
- Union Hospital affiliated to Tongji Medical College of Huazhong University of Science and Technology, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No